CLINICAL TRIAL: NCT05984615
Title: Real-world Evaluation of the Impact of Baseline Metastases on Clinical Outcomes Among BRAF Positive Metastatic Melanoma Patients
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CTMT212AUS63
Record Dates: First submitted 2023-08-02; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: BRAF Positive Metastatic Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Immunotherapy (IO) Cohort
- Targeted Therapy (TT) Cohort

SUMMARY:
This was a retrospective real-world evidence cohort study.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of melanoma (The International Classification of Diseases, 9th Revision [ICD-9] 172.x & 10th revision [ICD-10] C43 or D03x).
* Pathologic stage IV at initial diagnosis on or after 01 January 2011.
* First-line treatment with IO monotherapy or combination therapy (nivolumab, pembrolizumab, ipilimumab + nivolumab) or TT combination therapy (dabrafenib + trametinib, vemurafenib+cobimetinib, encorafenib+binimetinib) on or after 01 January 2014.
* Evidence of a BRAF test.
* Evidence of a BRAF-positive result prior to or up to 30 days after first-line (1L) therapy initiation.
* At least 18 years of age at the time of initiation of 1L treatment.

Exclusion criteria:

* Documented receipt of a clinical trial treatment for cancer at any time on or after 01 January 2014.
* Diagnosis of a second primary cancer or secondary cancer following initiation of 1L metastatic melanoma (MM) treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 1961 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-08-24 (Actual); Study Completion 2022-08-24 (Actual)

PRIMARY OUTCOMES:
Mean age | Baseline
Number of male patients | Baseline
Race | Baseline
Mean Charlson comorbidity index (CCI) score | Baseline
  Comorbidity was categorized into three grades: mild, with CCI scores of 1-2; moderate, with CCI scores of 3-4; and severe, with CCI scores ≥5.
Eastern Cooperative Oncology Group performance status (ECOG PS) | Baseline
  The ECOG scale consists of 4 grades (from 0 to 4) where 0 implies fully active, and 4 implies completely disabled.
Number of patients with study-related biomarkers | Baseline
  Study-related biomarkers included BRAF and PD1/PDL1 test dates and results.
Number of metastatic sites | Baseline

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 6 months and 1, 1.5, and 2 years
  PFS was defined as the time from the initiation of a line of therapy until the date of progression or death.
Overall survival (OS) | 6 months and 1, 1.5, and 2 years
  OS was defined as the time from the initiation of a line of therapy until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States